CLINICAL TRIAL: NCT07200830
Title: Radioligand Efficacy Comparison by Initial PSA-Response Outcome in Metastatic CRPC With Lutetium 177Lu PSMA RLT (RECIPROCAL)
Brief Title: Testing Different Dosing Schedules of the Anti-cancer Drug, Lutetium 177Lu PSMA RLT and Its Effect on Patients With Advanced Prostate Cancer, RECIPROCAL Trial
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A032304
Record Dates: First submitted 2025-09-23; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Castration-Resistant Prostate Carcinoma; Metastatic Prostate Adenocarcinoma; Stage IVB Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Pluvicto; Remote Patient Monitoring; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pre-registration step 0 (177Lu PSMA RLT) (Active Comparator): Patients receive 177Lu PSMA RLT IV on day 1 of each cycle. Cycles repeat every 6 weeks for up to 2 cycles in the absence of disease progression or unacceptable toxicity. Patients who achieve a PSA50 response at C2 D22 proceed to Step 1. Additionally, patients undergo blood sample collection, CT, and bone scan throughout the trial and PSMA PET during screening. Patients with a history of brain metastases or with clinical indication also undergo MRI throughout the trial.
  Interventions: Drug: Lutetium Lu 177 Vipivotide Tetraxetan; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Bone Scan; Procedure: PSMA PET Scan; Procedure: MRI; Other: Questionnaire Administration
- Randomization step 1 arm 1 (standard dose 177Lu PSMA RLT) (Active Comparator): Patients receive 177Lu PSMA RLT IV on day 1 of each cycle. Cycles repeat every 6 weeks for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo blood sample collection, CT, and bone scan throughout the trial and PSMA PET during screening. Patients with a history of brain metastases or with clinical indication also undergo MRI throughout the trial
  Interventions: Drug: Lutetium Lu 177 Vipivotide Tetraxetan; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Bone Scan; Procedure: PSMA PET Scan; Procedure: MRI; Other: Questionnaire Administration
- Randomization step 1 arm 2 (adaptive dose 177Lu PSMA RLT ) (Experimental): Starting cycle 2 day 42, patients undergo blood sample collection and PSA monitoring Q3W in the absence of disease progression or unacceptable toxicity. Patients with either an absolute PSA rise > 4 ng/dL, PSA rise > 25% above nadir, or clinical progression receive 177Lu PSMA RLT IV three weeks later. Patients then resume PSA monitoring Q3W with adaptive 177Lu PSMA RLT dosing as above for up to 4 total doses in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo blood sample collection, CT, and bone scan throughout the trial and PSMA PET during screening. Patients with a history of brain metastases or with clinical indication also undergo MRI throughout the trial.
  Interventions: Drug: Lutetium Lu 177 Vipivotide Tetraxetan; Procedure: Biospecimen Collection; Procedure: Patient Monitoring; Procedure: Computed Tomography; Procedure: Bone Scan; Procedure: PSMA PET Scan; Procedure: MRI; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Lutetium Lu 177 Vipivotide Tetraxetan — Given IV
  Other Names: Pluvicto
Procedure: Biospecimen Collection — Undergo blood sample collection
Procedure: Patient Monitoring — Undergo PSA monitoring
  Arms: Randomization step 1 arm 2 (adaptive dose 177Lu PSMA RLT )
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT Scan; CT Scan
Procedure: Bone Scan — Undergo Bone Scan
Procedure: PSMA PET Scan — Undergo PSMA PET Scan
Procedure: MRI — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This randomized phase III trial examines whether lengthening the dosage interval in an adaptive manner for the prostate cancer drug lutetium 177 Lu PSMA RLT improves quality of life without decreasing lifespan when compared to the standard way this medication is given. This study is for patients with hormone resistant prostate cancer that may have spread from where it first started to nearby tissue, lymph nodes, or distant parts of the body. Hormone resistant prostate cancer often has many cells containing a protein called prostate-specific membrane antigen (PSMA) on their surface. The normal cells in the prostate do not normally express as much PSMA protein on their surface as cancer cells. Lutetium 177 Lu PSMA RLT binds to the PSMA protein on the tumor cells. It builds up in these cells and gives off radiation that may kill them. Typically, this medication is given at the same dose every 6 weeks for up to 6 doses. In this trial, researchers want to see if treatment following the first two doses of lutetium 177 Lu PSMA RLT can be delayed until there is evidence of disease activity. This may be an effective way to improve quality of life without decreasing lifespan in patients with advanced prostate cancer.

DETAILED DESCRIPTION:
The primary and secondary objectives of the study:

PRIMARY OBJECTIVES:

I. To compare the overall survival (OS) of patients with metastatic castration-resistant prostate carcinoma (mCRPC) receiving prostate-specific antigen (PSA) adaptive dosing of lutetium 177 Lu prostate specific membrane antigen radioligand therapy (177Lu PSMA RLT) to that of patients receiving standard dose 177Lu PSMA RLT every 6 weeks.

II. To compare quality of life, as measured by Functional Assessment of Cancer Therapy- Prostate (FACT-P) total scores averaged across the first 30 months, in patients with mCRPC who receive 177Lu PSMA RLT adaptive dosing versus standard dosing.

SECONDARY OBJECTIVES:

I. To compare the duration of treatment between standard dosing and adaptive dosing.

II. To compare the radiographic progression-free survival (rPFS) between the treatment arms.

III. To evaluate and compare the toxicity profile of 177Lu PSMA RLT standard dosing and 177Lu PSMA RLT adaptive dosing.

IV. To compare the nadir PSA and PSA kinetics between standard and adaptive dosing.

V. To compare quality-adjusted life years, which accounts for overall survival and health utility (measured by European Quality of Life Five Dimension Five Level Scale [EQ-5D-5L]), between arms.

VI. To compare pain severity, as measured by the Brief Pain Inventory - Short Form (BPI-SF), between arms at 12 and 30 months.

EXPLORATORY OBJECTIVES:

I. To determine the frequency of tumor genomic aberrations (including but not limited to androgen receptor [AR] mutation/amplification, deoxyribonucleic acid [DNA] repair, retinoblastoma 1 [RB1], phosphatase and tensin homolog [PTEN], TP53) by circulating-tumor deoxyribonucleic acid (ctDNA) in patients achieving > 50% PSA decline versus (vs) < 50% PSA decline after 2 cycles of 177Lu PSMA RLT.

II. To evaluate the relationship between OS and initial PSA response (e.g. ≥ 50% decline in PSA level from baseline [PSA50] vs ≥ 75% decline in PSA level from baseline [PSA75] vs ≥ 90% decline in PSA level from baseline [PSA90]) prior to randomization.

OUTLINE:

PRE-REGISTRATION STEP 0: Patients receive 177Lu PSMA RLT intravenously (IV) on day 1 of each cycle. Cycles repeat every 6 weeks for up to 2 cycles in the absence of disease progression or unacceptable toxicity. Patients who achieve a PSA50 response at cycle (C) 2 day (D) 22 proceed to Step 1.

RANDOMIZATION STEP 1: Patients are randomized to 1 of 2 arms.

ARM 1: Patients receive 177Lu PSMA RLT IV on day 1 of each cycle. Cycles repeat every 6 weeks for up to 4 cycles in the absence of disease progression or unacceptable toxicity.

ARM 2: Starting cycle 2 day 42, patients undergo blood sample collection and PSA monitoring once every 3 weeks (Q3W) in the absence of disease progression or unacceptable toxicity. Patients with either an absolute PSA rise > 4 ng/dL, PSA rise > 25% above nadir, or clinical progression receive 177Lu PSMA RLT IV three weeks later. Patients then resume PSA monitoring Q3W with adaptive 177Lu PSMA RLT dosing for up to 4 total doses in the absence of disease progression or unacceptable toxicity.

Additionally, all patients undergo blood sample collection, computed tomography (CT), and bone scan throughout the trial and PSMA positron emission tomography (PET) during screening. Patients with a history of brain metastases or with clinical indication also undergo magnetic resonance imaging (MRI) throughout the trial.

After completion of study treatment, patients are followed up every 12 weeks until disease progression and then every 6 months thereafter for 5 years following registration.

ELIGIBILITY:
Inclusion Criteria:

* PRE-REGISTRATION (STEP 0): Patients must have histological, pathological, and/or cytological confirmation of prostate adenocarcinoma
* PRE-REGISTRATION (STEP 0): Patients must have a positive PSMA PET/CT scan (either gallium Ga 68 gozetotide [68Ga-PSMA-11], fluorine F 18 piflufolastat [18F- DCFPyl], or fluorine F 18 flotufolastat gallium [18F-rhPSMA-7.3]), as defined as uptake greater than liver with no PSMA negative measurable soft tissue disease
* PRE-REGISTRATION (STEP 0): PSA greater than 2.0 ng/mL
* PRE-REGISTRATION (STEP 0): Patients must have progressive mCRPC. Documented progressive mCRPC will be based on at least 1 of the following criteria:

  * Serum PSA progression defined as 2 consecutive increases in PSA over a previous reference value measured at least 1 week prior. The minimal start value is 2.0 ng/mL
  * Soft-tissue progression defined as an increase ≥ 20% in the sum of the diameter (SOD) (short axis for nodal lesions and long axis for non-nodal lesions) of all target lesions based on the smallest SOD since treatment started or the appearance of one or more new lesions
  * Progression of bone disease: evaluable disease or new bone lesions(s) by bone scan (2+2 Prostate Cancer Clinical Trials Working Group 3 [PCWG3] criteria, Scher et al 2016)
* PRE-REGISTRATION (STEP 0): Patients must have prior orchiectomy and/or ongoing androgen-deprivation therapy and a castrate level of serum testosterone (< 50 ng/dL or < 1.7 nmol/L)
* PRE-REGISTRATION (STEP 0): Patients must have received at least one androgen receptor pathway inhibitor (ARPI) (to include either apalutamide, darolutamide, enzalutamide, or abiraterone)

  * ARPI must be stopped at least 4 weeks prior to pre-registration
* PRE-REGISTRATION (STEP 0): Patients must not have previously received a taxane based chemotherapy regimen for mCRPC. Prior docetaxel for metastatic hormone-sensitive prostate carcinoma (mHSPC) or in the neoadjuvant or adjuvant setting is permitted if completed at least 12 months prior to pre-registration
* PRE-REGISTRATION (STEP 0): Patients must have recovered to ≤ grade 2 from all clinically significant toxicities related to prior therapies (i.e. prior chemotherapy, radiation, immunotherapy, etc.)
* PRE-REGISTRATION (STEP 0): Patients on a stable bisphosphonate or denosumab regimen for ≥ 30 days prior to pre-registration are eligible
* PRE-REGISTRATION (STEP 0): Previous treatment with strontium Sr-89 (strontium-89), samarium Sm-153 (samarium-153), rhenium Re 186 (rhenium-186), rhenium Re 188 (rhenium-188), radium Ra 223 (radium-223) or hemi-body irradiation within 6 months prior to pre-registration is not allowed. Previous PSMA-targeted radioligand therapy is not allowed
* PRE-REGISTRATION (STEP 0): Any systemic anti-cancer therapy (e.g. chemotherapy, immunotherapy or biological therapy [including monoclonal antibodies]) within 28 days prior to pre-registration is not allowed
* PRE-REGISTRATION (STEP 0): Age ≥ 18 years
* PRE-REGISTRATION (STEP 0): Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 2
* PRE-REGISTRATION (STEP 0): Absolute neutrophil count (ANC) ≥ 1,500/mm^3
* PRE-REGISTRATION (STEP 0): Platelet count ≥ 100,000/mm^3
* PRE-REGISTRATION (STEP 0): Total bilirubin < 1.5 x upper limit of normal (ULN) or < 3 x ULN in patients with Gilbert's syndrome
* PRE-REGISTRATION (STEP 0): Creatinine clearance estimated glomerular filtration rate (eGFR) ≥ 40 mL/min/1.73m^2 using the Modification of Diet in Renal Disease (MDRD) equation
* PRE-REGISTRATION (STEP 0): No acute biliary or urinary obstruction
* PRE-REGISTRATION (STEP 0): Patients with treated/stable brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression

  * Patients with a history of CNS metastases must have received therapy (surgery, radiotherapy, gamma knife) and be neurologically stable, asymptomatic, and not receiving corticosteroids for the purposes of maintaining neurologic integrity. Patients with epidural disease, canal disease and prior cord involvement are eligible if those areas have been treated, are stable, and not neurologically impaired. For patients with parenchymal CNS metastasis (or a history of CNS metastasis), baseline and subsequent radiological imaging must include evaluation of the brain (MRI preferred or CT with contrast)
* PRE-REGISTRATION (STEP 0): Patients with known HIV infection on effective anti-retroviral therapy with undetectable viral load within 6 months prior to registration are eligible for this trial
* PRE-REGISTRATION (STEP 0): For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* PRE-REGISTRATION (STEP 0): Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* PRE-REGISTRATION (STEP 0): Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class II or better
* PRE-REGISTRATION (STEP 0): No investigational agents within 28 days prior to pre-registration
* PRE-REGISTRATION (STEP 0): No other concurrent cytotoxic chemotherapy, immunotherapy, radioligand therapy, or investigational therapy
* PRE-REGISTRATION (STEP 0): No known hypersensitivity to the components of the study therapy or its analogs
* PRE-REGISTRATION (STEP 0): No transfusion within 30 days of pre-registration
* PRE-REGISTRATION (STEP 0): No symptomatic cord compression, or clinical or radiologic findings indicative of impending cord compression
* PRE-REGISTRATION (STEP 0): Ability to read and comprehend English or Spanish
* REGISTRATION (STEP 1): Completion of 2 doses of 177Lu PSMA RLT
* REGISTRATION (STEP 1): PSA decline ≥ 50% between C1 D1 (screening) and C2 D22 +/-3 days
* REGISTRATION (STEP 1): ECOG Performance Status ≤ 2
* REGISTRATION (STEP 1): Absolute neutrophil count (ANC) ≥ 1,500/mm^3
* REGISTRATION (STEP 1): Platelet count ≥ 100,000/mm^3
* REGISTRATION (STEP 1): Creatinine clearance eGFR ≥ 40 mL/min/1.73m^2 using the Modification of Diet in Renal Disease (MDRD) equation

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1524 (Estimated)
Dates: Start 2025-10-08 (Estimated); Primary Completion 2034-09-09 (Estimated); Study Completion 2034-09-09 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | Up to 5 years
  Will be calculated as time from randomization until death due to any cause, censoring patients not known to have died at the time of their last follow-up. OS will be compared between the treatment arms using a stratified log rank test
Quality of life | Up to 30 months
  Will be measured using the Functional Assessment of Cancer Therapy- Prostate (FACT-P) total scores. A repeated measures mixed model will be used to evaluate the between-arm mean difference in FACT-P Total scores across the first 30 months from treatment start. A point estimate of the difference and 95% confidence interval will be reported. Results of formal hypothesis testing will only be reported if adaptive dosing is deemed noninferior to standard dosing with regards to overall survival.

SECONDARY OUTCOMES:
Duration of treatment | Up to 5 years
  Calculated from the first administration of 177Lu PSMA RLT to the last administration of 177Lu PSMA RLT among randomized patients. Summary measures for the duration of treatment will be recorded by arm and the stratified Wilcoxon rank sum statistic will be used to test whether the treatment duration distribution differs between the standard and adaptive dose treatments.
Radiographic progression-free survival (rPFS) | Up to 5 years
  Will be defined as time from randomization to the to the date of radiographic disease progression per the Prostate Cancer Clinical Trials Working Group 3 criteria or death from any cause, whichever occurs first. Patients who are alive without a disease progression will be censored at the time of their last disease evaluation. rPFS will be compared between the two treatment arms using a stratified logrank test.
Rate of Grade 3+ AEs | Up to 5 years
  Will be assessed using Common Terminology Criteria for Adverse Events version 5.0. The proportion of patients that experience a grade 3+ AE regardless of attribution will be summarized as the number and percent of patients by treatment arm.
Prostate-specific antigen (PSA) response | Prior to randomization
  There will be different thresholds used for PSA response, all measured as change from baseline and confirmed at least 3 weeks later by a second PSA test: PSA50 (a ≥ 50% decline), PSA75 (a ≥ 75% decline), and PSA90 (a ≥ 90% decline).
Nadir PSA | Up to 5 years
  This is the lowest PSA value observed starting from baseline.
Pain Severity | Up to 30 months
  This will be measured using the Brief Pain Index Short Form (BPI-SF). Estimates and 95% confidence intervals for the mean difference between treatment arms at 12 and 30 months will be generated using a repeated measures mixed model.
Quality-adjusted life years | Up to 5 years
  This will be calculated from overall survival and health utility as measured by European Quality of Life Five Dimension Five Level Scale (EQ-5D-5L) using an area under the curve approach. Summary statistics for the area under the curve of each arm and a 95% CI for the difference between arms will be reported.

OTHER OUTCOMES:
Frequency of tumor genomic aberrations | Up to 3 months
  : Investigated tumor genomic aberrations include androgen receptor mutation/amplification, deoxyribonucleic acid repair, retinoblastoma 1, phosphatase and tensin homolog, and TP53. The frequency will be compared between treatment arms using a two-sample t-test (or a Fisher's exact test if more appropriate) among patients with ≥ 50% PSA decline and < 50% PSA decline after 2 cycles of 177Lu PSMA RLT.
Association between initial PSA response and OS | Up to 5 years
  The median survival time will be computed by the Kaplan-Meier estimator for patients with a pre-randomization PSA response between ≥ 50% and < 75%, ≥ 75% and less than 90%, and ≥ 90%. A log rank test will be used to compare OS between the three groups.
Estimate of treatment effect by race | up to 5 years
  Estimates of the OS HR and the corresponding 95% CIs by race
Estimate of treatment effect by ethnicity | up to 5 years
  Estimates of the OS HR and the corresponding 95% CIs by ethnicity

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Hope, MD, Study Chair — Alliance for Clinical Trials in Oncology

IPD SHARING:
Plan to Share IPD: Undecided